CLINICAL TRIAL: NCT00305097
Title: Effects of Caffeinated and Decaffeinated Coffee on Body Weight and Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Harvard School of Public Health (HSPH) (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DK46200 (completed); P30DK046200 (NIH)
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Overweight
Keywords: coffee; caffeine; glucose tolerance; body weight; insulin sensitivity; randomized controlled trial
MeSH Terms: conditions — Overweight; Body Weight; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caffeinated coffee (Experimental): Caffeinated coffee
  Interventions: Dietary Supplement: Caffeinated coffee
- Decaffeinated coffee (Experimental): Decaffeinated coffee
  Interventions: Dietary Supplement: Decaffeinated coffee
- No coffee (Active Comparator)
  Interventions: Dietary Supplement: No coffee

INTERVENTIONS:
Dietary Supplement: Decaffeinated coffee — 5 cups per day for 8 weeks
  Other Names: Instant Nestle decaffeinated coffee
  Arms: Decaffeinated coffee
Dietary Supplement: Caffeinated coffee — 5 cups per day for 8 weeks
  Other Names: Instant Nestle caffeinated coffee
  Arms: Caffeinated coffee
Dietary Supplement: No coffee
  Arms: No coffee

SUMMARY:
Habitual consumption of coffee may have substantial beneficial effects on glucose metabolism according to recent findings of epidemiological studies in the U.S., Europe, and Japan. However, data from longer-term human intervention studies with appropriate outcome measures are lacking. We will study the effects of caffeinated and decaffeinated coffee consumption on body fatness, insulin sensitivity and glucose tolerance that may underlie the observed associations with a lower risk of type 2 diabetes in a randomized controlled trial. We hypothesize that both caffeinated and decaffeinated coffee will improve insulin sensitivity and glucose tolerance. Before starting a larger, long-term intervention study, we will conduct a pilot study to test the feasibility of such a trial. The pilot study will be an 8-week parallel trial in 45 overweight individuals, who will be randomized to drinking 5 cups per day of 1) caffeinated coffee (n=15), 2) decaffeinated coffee (n=15), or 3) water (n=15). Body fatness (weight, waist circumference, bioelectrical impedance), insulin sensitivity (HOMA model), and glucose tolerance (oral glucose tolerance test) will be the primary outcomes. We will assess the adherence of participants to their assigned treatment by measuring serum caffeine concentrations, documentation of coffee use in diaries by the participants, and counting unused coffee packets. We will also obtain feedback from participants on how to improve compliance in a future trial. If successful, this study will form the basis for a definitive trial of coffee consumption, body fatness, and glucose tolerance. Given the extensive use of coffee and the rapidly increasing health burden of type 2 diabetes, such a trial would have important public health implications.

DETAILED DESCRIPTION:
Habitual consumption of coffee may have substantial beneficial effects on glucose metabolism according to recent findings of epidemiological studies in the U.S., Europe, and Japan. However, data from longer-term human intervention studies with appropriate outcome measures are lacking. We will study the effects of caffeinated and decaffeinated coffee consumption on body fatness, insulin sensitivity and glucose tolerance that may underlie the observed associations with a lower risk of type 2 diabetes in a randomized controlled trial. We hypothesize that both caffeinated and decaffeinated coffee will improve insulin sensitivity and glucose tolerance. Before starting a larger, long-term intervention study, we will conduct a pilot study to test the feasibility of such a trial. The pilot study will be an 8-week parallel trial in 45 overweight individuals, who will be randomized to drinking 5 cups per day of 1) caffeinated coffee (n=15), 2) decaffeinated coffee (n=15), or 3) water (n=15). Body fatness (weight, waist circumference, bioelectrical impedance), insulin sensitivity (HOMA model), and glucose tolerance (oral glucose tolerance test) will be the primary outcomes. We will assess the adherence of participants to their assigned treatment by measuring serum caffeine concentrations, documentation of coffee use in diaries by the participants, and counting unused coffee packets. We will also obtain feedback from participants on how to improve compliance in a future trial. If successful, this study will form the basis for a definitive trial of coffee consumption, body fatness, and glucose tolerance. Given the extensive use of coffee and the rapidly increasing health burden of type 2 diabetes, such a trial would have important public health implications.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years with an ability and willingness to give written informed consent.
* Body mass index 25-35 kg/m2
* Users of at least 2 cups of caffeinated coffee per day who are willing to be randomized to any of the interventions.
* Non-smoking

Exclusion Criteria:

* Any condition/illness that may affect the study outcomes or would make participation potentially harmful such as pregnancy or breastfeeding, diabetes mellitus, heart disease, stroke, hypertension, malabsorption syndromes, Gastroesophageal reflux disease GERD, a history of ulcer, according to a detailed medical history.
* Abnormal hepatic function (liver function test > twice the normal range), abnormal renal function (creatinine > 1.1 mg/dl), fasting plasma glucose in the diabetic range (>/= 126 mg/dl), or blood pressure > 140/90 mmHg.
* Present alcoholism or drug abuse or use of medications that could interfere with the treatment including bronchodilators, quinolone antibiotics, monoamine oxidase inhibitors, anxiolytics, ranitidine, corticosteroids, growth hormone, antihypertensives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
glucose tolerance / insulin sensitivity | 4 and 8 weeks

SECONDARY OUTCOMES:
body weight/fatness, blood pressure, concentrations of blood lipids, adipokines, inflammatory markers | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rob M van Dam, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Christos Mantzoros, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Wedick NM, Brennan AM, Sun Q, Hu FB, Mantzoros CS, van Dam RM. Effects of caffeinated and decaffeinated coffee on biological risk factors for type 2 diabetes: a randomized controlled trial. Nutr J. 2011 Sep 13;10:93. doi: 10.1186/1475-2891-10-93. PMID 21914162
- [Derived] Peter PR, Park KH, Huh JY, Wedick NM, Mantzoros CS. Circulating irisin levels are not affected by coffee intake: a randomized controlled trial. PLoS One. 2014 Apr 11;9(4):e94463. doi: 10.1371/journal.pone.0094463. eCollection 2014. PMID 24728416
- [Derived] Wedick NM, Mantzoros CS, Ding EL, Brennan AM, Rosner B, Rimm EB, Hu FB, van Dam RM. The effects of caffeinated and decaffeinated coffee on sex hormone-binding globulin and endogenous sex hormone levels: a randomized controlled trial. Nutr J. 2012 Oct 19;11:86. doi: 10.1186/1475-2891-11-86. PMID 23078574